CLINICAL TRIAL: NCT00600301
Title: Vitrectomy Without Internal Limiting Membrane Removal in the Treatment of Diffuse Diabetic Macular Edema: a Comparative Kenalog Vs Bevacizumab Intravitreal Injection Vs Control Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-OO13
Record Dates: First submitted 2006-06-30; First posted 2008-01-24 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Diffuse Diabetic Macular Edema
Keywords: Macula; Edema
MeSH Terms: conditions — Edema | interventions — Triamcinolone Acetonide; Bevacizumab

INTERVENTIONS:
Drug: Triamcinolone Acetonide and Bevacizumab

SUMMARY:
Diabetic macular edema is the most common cause of visual loss among patients with diabetic retinopathy. Pars plana vitrectomy has been reported to be effective for the treatment of diabetic macular edema. Previous report showed a limited improvement in visual acuity and macular thickness posterior intraoperative triamcinolone acetonide. Bevacizumab intravitreal injection has been proven be effective in the treatment of diabetic macular edema, in recent publications. The purpose of this study is to evaluate whether vitrectomy with and without intravitreal triamcinolone acetonide and bevacizumab injection affects vision outcome and macular thickness in patients with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse diabetic macular edema
* Non proliferative diabetic retinopathy
* No VPP previa
* No previous treament with laser, Triamcinolone acetonide, and Bevacizumab

Exclusion Criteria:

* Proliferative diabetic retinopathy
* Previous pars plana vitrectomy
* Previous treatment with diabetic macular edema
* Focal macular edema
* Macular Ischemia

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maximiliano Gordon, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociacion Para Evitar la Ceguera en Mexico, México, Mexico